CLINICAL TRIAL: NCT03462030
Title: Phase II Study of Baked Milk Oral Immunotherapy for the Treatment of Cow's Milk Allergy
Brief Title: Baked Milk Oral Immunotherapy for Cow's Milk Allergy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Myra Reinhardt Foundation (Other); La Jolla Institute for Allergy & Immunology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00099590
Record Dates: First submitted 2018-02-28; First posted 2018-03-12 (Actual); Results first posted 2021-12-03 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Cow's Milk Allergy
Keywords: food allergy; oral immunotherapy
MeSH Terms: conditions — Milk Hypersensitivity; Food Hypersensitivity | interventions — Drugs, Investigational

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Baked Milk Immunotherapy (Experimental): Subjects will receive baked milk oral immunotherapy with baked non-fat cow's milk powder as the intervention. Subjects will undergo an initial dose escalation, build-up, and then a maintenance period.
  Interventions: Drug: Baked non-fat cow's milk powder
- Placebo (Placebo Comparator): Subjects will receive oral immunotherapy with the placebo control (tapioca powder). Subjects will undergo an initial dose escalation, build-up, and then a maintenance period.
  Interventions: Drug: Placebo: Tapioca Powder

INTERVENTIONS:
Drug: Baked non-fat cow's milk powder — Oral immunotherapy with increasing quantities of baked milk.
  Other Names: Investigational New Drug (IND) 17114
  Arms: Baked Milk Immunotherapy
Drug: Placebo: Tapioca Powder — Placebo control.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether baked milk oral immunotherapy is safe in the treatment of cow's milk allergy.

DETAILED DESCRIPTION:
This study is designed to assess the safety of baked milk oral immunotherapy among patients who are milk allergic and who do not pass a baked milk challenge.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet all of the following criteria are eligible for enrollment as study participants, including participants who:

  * Are age 3-18 years, either sex, any ethnicity or race
  * Provide signed informed consent by parent or legal guardian and informed assent if applicable
  * Have a history of symptomatic reactivity to cow's milk (i.e. eczema, urticarial, upper or lower respiratory symptoms, gastrointestinal disturbances, rash, oral symptoms)
  * Have a skin prick test positive to milk (diameter of wheal 3 mm ≥ negative control) and serum milk-specific immunoglobulin E (IgE) level >5 kilo Units (kU)/L within the past 6-12 months
  * Have a positive reaction to a cumulative dose of ≤444 mg of baked milk powder in the initial qualifying double blind placebo-controlled food challenge.
  * Use an effective method of contraception by females of childbearing potential to prevent pregnancy and agree to continue to practice an acceptable method of contraception for the duration of their participation in the study.
  * Have self-injectable epinephrine available at all times

Exclusion Criteria:

* Patients who meet any of these criteria are not eligible for enrollment as study participants, including participants who:

  * Have a history of severe anaphylaxis resulting in hypotension, neurological compromise, or mechanical ventilation
  * Have a history of intubation related to asthma
  * Tolerate more than 444 mg of baked milk powder at the initial qualifying double blind placebo controlled food challenge.
  * Allergy to placebo ingredients or reacts to any dose of placebo during the qualifying oral food challenge.
  * Poor control of atopic dermatitis
  * Are unable to tolerate at least 3 mg of baked milk protein on dose escalation day
  * Are pregnant or lactating
  * Have severe asthma defined by 2007 National Heart Lung and Blood Institute (NHLBI) Criteria Steps 5 or 6
  * Have severe or poorly controlled asthma defined by with any of the following criteria:

    1. Forced expiratory volume in 1 second (FEV1) <80% of predicted
    2. Inhaled corticosteroid dosing dosing of >500 mcg daily of fluticasone (or equivalent inhaled corticosteroids based on NHLBI dosing chart) or
    3. ≥ 1 hospitalization in the past year for asthma or
    4. > 1 emergency department visit in the past 6 months for asthma
  * Use of steroid medications (oral steroids, such as prednisone or Medrol, steroid injections, such as Kenalog, or intravenous or oral corticosteroid burst) in the following manners: History of daily oral steroid dosing within 4 weeks prior to baseline visit or for > 1 month during the past year or >2 burst oral steroid courses in the past 6 months.
  * Are unable to discontinue antihistamines for 5 days for long acting and 3 days for short acting prior to skin testing or food challenges
  * Are receiving omalizumab, mepolizumab, beta- blocker, angiotensin-converting-enzyme inhibitor (ACE-I), angiotensin-receptor blockers, calcium channel blockers, or tricyclic antidepressant therapy
  * Have used immunomodulatory therapy (not including corticosteroids) or biologic therapy within the past year
  * Have participated in any interventional study for treatment of a food allergy in the past 6 months
  * Are on 'build up phase' of environmental allergen immunotherapy. Subjects tolerating maintenance allergen immunotherapy can be enrolled.
  * Have a history of eosinophilic esophagitis in the past 3 years
  * Have a chronic disease (other than asthma, atopic dermatitis, rhinitis) requiring therapy (e.g., heart disease, diabetes)
  * Have used an investigational drug within 90 days or plan to use an investigational drug during the study period
  * Severe reaction at initial double blind placebo controlled food challenge, defined as:

    * Life-threatening anaphylaxis
    * Requiring overnight hospitalization

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2024-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wood, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Boyce JA, Assa'ad A, Burks AW, Jones SM, Sampson HA, Wood RA, Plaut M, Cooper SF, Fenton MJ, Arshad SH, Bahna SL, Beck LA, Byrd-Bredbenner C, Camargo CA Jr, Eichenfield L, Furuta GT, Hanifin JM, Jones C, Kraft M, Levy BD, Lieberman P, Luccioli S, McCall KM, Schneider LC, Simon RA, Simons FE, Teach SJ, Yawn BP, Schwaninger JM. Guidelines for the diagnosis and management of food allergy in the United States: summary of the NIAID-sponsored expert panel report. Nutr Res. 2011 Jan;31(1):61-75. doi: 10.1016/j.nutres.2011.01.001. No abstract available. PMID 21310308
- [Background] Gupta RS, Springston EE, Warrier MR, Smith B, Kumar R, Pongracic J, Holl JL. The prevalence, severity, and distribution of childhood food allergy in the United States. Pediatrics. 2011 Jul;128(1):e9-17. doi: 10.1542/peds.2011-0204. Epub 2011 Jun 20. PMID 21690110
- [Background] Chafen JJ, Newberry SJ, Riedl MA, Bravata DM, Maglione M, Suttorp MJ, Sundaram V, Paige NM, Towfigh A, Hulley BJ, Shekelle PG. Diagnosing and managing common food allergies: a systematic review. JAMA. 2010 May 12;303(18):1848-56. doi: 10.1001/jama.2010.582. PMID 20460624
- [Background] Sicherer SH, Sampson HA. Food allergy: Epidemiology, pathogenesis, diagnosis, and treatment. J Allergy Clin Immunol. 2014 Feb;133(2):291-307; quiz 308. doi: 10.1016/j.jaci.2013.11.020. Epub 2013 Dec 31. PMID 24388012
- [Background] Skripak JM, Matsui EC, Mudd K, Wood RA. The natural history of IgE-mediated cow's milk allergy. J Allergy Clin Immunol. 2007 Nov;120(5):1172-7. doi: 10.1016/j.jaci.2007.08.023. Epub 2007 Nov 1. PMID 17935766
- [Background] Wood RA, Sicherer SH, Vickery BP, Jones SM, Liu AH, Fleischer DM, Henning AK, Mayer L, Burks AW, Grishin A, Stablein D, Sampson HA. The natural history of milk allergy in an observational cohort. J Allergy Clin Immunol. 2013 Mar;131(3):805-12. doi: 10.1016/j.jaci.2012.10.060. Epub 2012 Dec 28. PMID 23273958
- [Background] Kim J, Kwon J, Noh G, Lee SS. The effects of elimination diet on nutritional status in subjects with atopic dermatitis. Nutr Res Pract. 2013 Dec;7(6):488-94. doi: 10.4162/nrp.2013.7.6.488. Epub 2013 Nov 29. PMID 24353835
- [Background] Hobbs CB, Skinner AC, Burks AW, Vickery BP. Food allergies affect growth in children. J Allergy Clin Immunol Pract. 2015 Jan-Feb;3(1):133-4.e1. doi: 10.1016/j.jaip.2014.11.004. Epub 2014 Nov 25. PMID 25577638
- [Background] Cummings AJ, Knibb RC, King RM, Lucas JS. The psychosocial impact of food allergy and food hypersensitivity in children, adolescents and their families: a review. Allergy. 2010 Aug;65(8):933-45. doi: 10.1111/j.1398-9995.2010.02342.x. Epub 2010 Feb 22. PMID 20180792
- [Background] Flokstra-de Blok BM, Dubois AE, Vlieg-Boerstra BJ, Oude Elberink JN, Raat H, DunnGalvin A, Hourihane JO, Duiverman EJ. Health-related quality of life of food allergic patients: comparison with the general population and other diseases. Allergy. 2010 Feb;65(2):238-44. doi: 10.1111/j.1398-9995.2009.02121.x. Epub 2009 Oct 1. PMID 19796214
- [Background] Eigenmann PA, Caubet JC, Zamora SA. Continuing food-avoidance diets after negative food challenges. Pediatr Allergy Immunol. 2006 Dec;17(8):601-5. doi: 10.1111/j.1399-3038.2006.00455.x. PMID 17121588
- [Background] Burbank AJ, Sood P, Vickery BP, Wood RA. Oral Immunotherapy for Food Allergy. Immunol Allergy Clin North Am. 2016 Feb;36(1):55-69. doi: 10.1016/j.iac.2015.08.007. PMID 26617227
- [Background] Nowak-Wegrzyn A, Bloom KA, Sicherer SH, Shreffler WG, Noone S, Wanich N, Sampson HA. Tolerance to extensively heated milk in children with cow's milk allergy. J Allergy Clin Immunol. 2008 Aug;122(2):342-7, 347.e1-2. doi: 10.1016/j.jaci.2008.05.043. Epub 2008 Jul 11. PMID 18620743
- [Background] Kim JS, Nowak-Wegrzyn A, Sicherer SH, Noone S, Moshier EL, Sampson HA. Dietary baked milk accelerates the resolution of cow's milk allergy in children. J Allergy Clin Immunol. 2011 Jul;128(1):125-131.e2. doi: 10.1016/j.jaci.2011.04.036. Epub 2011 May 23. PMID 21601913
- [Background] Oppenheimer JJ, Nelson HS, Bock SA, Christensen F, Leung DY. Treatment of peanut allergy with rush immunotherapy. J Allergy Clin Immunol. 1992 Aug;90(2):256-62. doi: 10.1016/0091-6749(92)90080-l. PMID 1500630
- [Background] Nelson HS, Lahr J, Rule R, Bock A, Leung D. Treatment of anaphylactic sensitivity to peanuts by immunotherapy with injections of aqueous peanut extract. J Allergy Clin Immunol. 1997 Jun;99(6 Pt 1):744-51. doi: 10.1016/s0091-6749(97)80006-1. PMID 9215240
- [Background] Hofmann AM, Scurlock AM, Jones SM, Palmer KP, Lokhnygina Y, Steele PH, Kamilaris J, Burks AW. Safety of a peanut oral immunotherapy protocol in children with peanut allergy. J Allergy Clin Immunol. 2009 Aug;124(2):286-91, 291.e1-6. doi: 10.1016/j.jaci.2009.03.045. Epub 2009 May 27. PMID 19477496
- [Background] Keet CA, Frischmeyer-Guerrerio PA, Thyagarajan A, Schroeder JT, Hamilton RG, Boden S, Steele P, Driggers S, Burks AW, Wood RA. The safety and efficacy of sublingual and oral immunotherapy for milk allergy. J Allergy Clin Immunol. 2012 Feb;129(2):448-55, 455.e1-5. doi: 10.1016/j.jaci.2011.10.023. Epub 2011 Nov 30. PMID 22130425
- [Background] Martorell A, De la Hoz B, Ibanez MD, Bone J, Terrados MS, Michavila A, Plaza AM, Alonso E, Garde J, Nevot S, Echeverria L, Santana C, Cerda JC, Escudero C, Guallar I, Piquer M, Zapatero L, Ferre L, Bracamonte T, Muriel A, Martinez MI, Felix R. Oral desensitization as a useful treatment in 2-year-old children with cow's milk allergy. Clin Exp Allergy. 2011 Sep;41(9):1297-304. doi: 10.1111/j.1365-2222.2011.03749.x. Epub 2011 Apr 11. PMID 21481024
- [Background] Meglio P, Bartone E, Plantamura M, Arabito E, Giampietro PG. A protocol for oral desensitization in children with IgE-mediated cow's milk allergy. Allergy. 2004 Sep;59(9):980-7. doi: 10.1111/j.1398-9995.2004.00542.x. PMID 15291907
- [Background] Longo G, Barbi E, Berti I, Meneghetti R, Pittalis A, Ronfani L, Ventura A. Specific oral tolerance induction in children with very severe cow's milk-induced reactions. J Allergy Clin Immunol. 2008 Feb;121(2):343-7. doi: 10.1016/j.jaci.2007.10.029. Epub 2007 Dec 26. PMID 18158176
- [Background] Skripak JM, Nash SD, Rowley H, Brereton NH, Oh S, Hamilton RG, Matsui EC, Burks AW, Wood RA. A randomized, double-blind, placebo-controlled study of milk oral immunotherapy for cow's milk allergy. J Allergy Clin Immunol. 2008 Dec;122(6):1154-60. doi: 10.1016/j.jaci.2008.09.030. Epub 2008 Oct 25. PMID 18951617
- [Background] Narisety SD, Skripak JM, Steele P, Hamilton RG, Matsui EC, Burks AW, Wood RA. Open-label maintenance after milk oral immunotherapy for IgE-mediated cow's milk allergy. J Allergy Clin Immunol. 2009 Sep;124(3):610-2. doi: 10.1016/j.jaci.2009.06.025. Epub 2009 Aug 8. PMID 19665770
- [Background] Pajno GB, Caminiti L, Ruggeri P, De Luca R, Vita D, La Rosa M, Passalacqua G. Oral immunotherapy for cow's milk allergy with a weekly up-dosing regimen: a randomized single-blind controlled study. Ann Allergy Asthma Immunol. 2010 Nov;105(5):376-81. doi: 10.1016/j.anai.2010.03.015. Epub 2010 Jul 31. PMID 21055664
- [Background] Yeung JP, Kloda LA, McDevitt J, Ben-Shoshan M, Alizadehfar R. Oral immunotherapy for milk allergy. Cochrane Database Syst Rev. 2012 Nov 14;11(11):CD009542. doi: 10.1002/14651858.CD009542.pub2. PMID 23152278
- [Background] Wood RA. Food allergen immunotherapy: Current status and prospects for the future. J Allergy Clin Immunol. 2016 Apr;137(4):973-982. doi: 10.1016/j.jaci.2016.01.001. PMID 27059725
- [Background] Wood RA, Kim JS, Lindblad R, Nadeau K, Henning AK, Dawson P, Plaut M, Sampson HA. A randomized, double-blind, placebo-controlled study of omalizumab combined with oral immunotherapy for the treatment of cow's milk allergy. J Allergy Clin Immunol. 2016 Apr;137(4):1103-1110.e11. doi: 10.1016/j.jaci.2015.10.005. Epub 2015 Nov 12. PMID 26581915
- [Background] Goldberg MR, Nachshon L, Appel MY, Elizur A, Levy MB, Eisenberg E, Sampson HA, Katz Y. Efficacy of baked milk oral immunotherapy in baked milk-reactive allergic patients. J Allergy Clin Immunol. 2015 Dec;136(6):1601-1606. doi: 10.1016/j.jaci.2015.05.040. Epub 2015 Jul 17. PMID 26194541
- [Background] Lin MS, Tanner E, Lynn J, Friday GA Jr. Nonfatal systemic allergic reactions induced by skin testing and immunotherapy. Ann Allergy. 1993 Dec;71(6):557-62. PMID 8267250
- [Background] Devenney I, Falth-Magnusson K. Skin prick tests may give generalized allergic reactions in infants. Ann Allergy Asthma Immunol. 2000 Dec;85(6 Pt 1):457-60. doi: 10.1016/S1081-1206(10)62571-9. PMID 11152165
- [Background] Valyasevi MA, Maddox DE, Li JT. Systemic reactions to allergy skin tests. Ann Allergy Asthma Immunol. 1999 Aug;83(2):132-6. doi: 10.1016/S1081-1206(10)62624-5. PMID 10480586
- [Background] Bernstein DI, Wanner M, Borish L, Liss GM; Immunotherapy Committee, American Academy of Allergy, Asthma and Immunology. Twelve-year survey of fatal reactions to allergen injections and skin testing: 1990-2001. J Allergy Clin Immunol. 2004 Jun;113(6):1129-36. doi: 10.1016/j.jaci.2004.02.006. PMID 15208595
- [Derived] Dantzer JA, Lewis SA, Psoter KJ, Sutherland A, Frazier A, Richardson E, Maiche S, Seumois G, Peters B, Wood RA. Clinical and immunological outcomes after randomized trial of baked milk oral immunotherapy for milk allergy. JCI Insight. 2025 Jan 9;10(1):e184301. doi: 10.1172/jci.insight.184301. PMID 39782691

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Johns Hopkins (JH) Pediatric Allergy Clinic, Baltimore, MD from March 2018 to October 2019.
Pre-assignment Details: 41 subjects were consented and screened. Eleven (27%) did not have dose-limiting symptoms in their screening food challenge to 444mg of baked milk protein and were therefore ineligible for the study. 30 subjects were randomized 1:1.
Period: Overall Study
Arm/Group | Baked Milk Immunotherapy | Placebo
Started | 15 | 15
End of Build-up | 14 | 14
Month 12 Food Challenge | 14 | 14
Completed | 14 | 14
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Baked Milk Immunotherapy | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 15 | 27
  Between 18 and 65 years | 3 | 0 | 3
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 13 [4 to 18] | 7 [3 to 14] | 11 [3 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 7 | 9 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 15 | 14 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 12 | 9 | 21
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30
Cow's Milk IgE [Median (Full Range); unit: kU/L] — Cow's Milk IgE (kU/L) at baseline.
  kU/L | 114 [7 to 1625] | 87 [22 to 772] | 88 [7 to 1625]
Age at Milk Allergy Diagnosis [Median (Full Range); unit: months] | 8 [4 to 14] | 9 [4 to 24] | 8.5 [4 to 24]
Participants with Prior Baked Milk Exposure [Count of Participants; unit: Participants] | 12 | 10 | 22
Participants with a History of milk reaction [Count of Participants; unit: Participants]
  Unheated Milk Only | 3 | 5 | 8
  Baked Milk Only | 3 | 0 | 3
  Both Unheated and Baked Milk | 9 | 10 | 19
Current Atopic History [Count of Participants; unit: Participants]
  Asthma | 11 | 9 | 20
  Atopic dermatitis | 8 | 8 | 16
  Allergic rhinitis | 10 | 11 | 21
  Non-milk food allergies | 12 | 14 | 26
Alpha lactalbumin IgE (kU/L) [Median (Full Range); unit: kU/L] | 20.4 [0.6 to 556] | 19.7 [0.2 to 291] | 20 [0.2 to 556]
Beta lactoglobulin igE (kU/L) [Median (Full Range); unit: kU/L] | 28.2 [0.4 to 487] | 18.8 [4.1 to 79.3] | 24.5 [0.4 to 487]
Casein IgE (kU/L) [Median (Full Range); unit: kU/L] | 75.8 [5.9 to 1326] | 52.8 [15.4 to 652] | 64.8 [5.9 to 1326]
Milk IgG4 (mg/L) [Median (Full Range); unit: mg/L] | 8.6 [6.9 to 12.5] | 9.4 [7.4 to 19] | 9.2 [6.9 to 19]
Milk skin prick test [Median (Full Range); unit: mm] — Milk skin prick test (wheal size/diameter) measured in millimeters (mm).
  mm | 14 [7 to 23] | 10 [5 to 25] | 13 [5 to 25]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0
Description: Adverse events will be recorded per CTCAE version 4.0. Events per dose on baked milk oral immunotherapy will be compared to adverse events per dose on placebo. Data will be collected over the first year of treatment. Analysis of cumulative adverse reactions per dose of oral immunotherapy or placebo will be performed at the end of year 1.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Baked Milk Immunotherapy | Placebo
Number analyzed (Participants) | 15 | 15
Participants | 15 | 11

2. Secondary Outcome: Proportion of Subjects Who Are Able to Tolerate 4 Grams of Baked Milk Protein After One Year of Treatment
Description: The investigators will perform baked milk challenges to 4044 mg of baked milk protein and calculate the proportion of subjects who tolerate 4 grams of baked milk protein after one year of baked milk oral immunotherapy. This measure reports the number of participants that were able to tolerate 4 grams of baked milk protein.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Baked Milk Immunotherapy | Placebo
Number analyzed (Participants) | 15 | 15
Participants | 11 | 0

3. Secondary Outcome: Number of Subjects Who Are Able to Tolerate 2 Grams of Unheated Milk Protein After 2 Years of Treatment
Description: The investigators will perform unheated milk challenges to up to 8000 mg of unheated milk protein and calculate the proportion of subjects who tolerate 2 grams of unheated milk protein after 2 years of treatment. This measure reports the number of participants that were able to tolerate 2 grams of unheated milk protein.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Baked Milk Immunotherapy | Placebo
Number analyzed (Participants) | 15 | 15
Participants | 8 | 5

4. Secondary Outcome: Change in Maximum Tolerated Dose of Baked Milk
Description: Change in maximum tolerated dose (milligrams) of baked milk from baseline to end of year 1 and end of year 2.
Time Frame: Baseline, 1 year and 2 years
Measure: Median (95% Confidence Interval); unit: miligrams
Arm/Group | Baked Milk Immunotherapy | Placebo
Number analyzed (Participants) | 15 | 15
miligrams
  Change from baseline to 1 year | 3900 [2256 to 4025] | 0 [0 to 757]
  Change from baseline to 2 years | 3900 [2371 to 4025] | 3900 [2031 to 3900]

5. Secondary Outcome: Change in Milk-specific IgE Level
Description: Change in milk-specific immunoglobulin E (IgE) level measured in kU/L.
Time Frame: Baseline and up to year 2
Population: For change from baseline to year 1, 1 participant dropped out in each group so blood/results only available for 14 participants in each group. 4 participants dropped out in year 2 so blood/results was available for 12 in each group for change from baseline to year 2.
Measure: Median (95% Confidence Interval); unit: KU/L
Arm/Group | Baked Milk Immunotherapy | Placebo
Number analyzed (Participants) | 14 | 14
KU/L
  change from baseline to 1 year | -21.35 [-40.08 to 6.67] | -14.75 [-41.73 to 12.42]
  change from baseline to 2 years: number analyzed (Participants) | 12 | 12
  change from baseline to 2 years | -77.45 [-138.95 to -15.69] | -46.65 [-109.47 to -14.60]

6. Secondary Outcome: Change in Milk-specific IgG4 Level
Description: Change in milk-specific immunoglobulin G4 (IgG4) level measured in mg/L.
Time Frame: Baseline and up to year 2
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: mg/L
Arm/Group | Baked Milk Immunotherapy | Placebo
Number analyzed (Participants) | 14 | 14
mg/L
  change from baseline to 1 year | 8.88 [4.58 to 85.34] | 3.79 [2.69 to 4.26]
  Change from baseline to 2 years: number analyzed (Participants) | 12 | 12
  Change from baseline to 2 years | 5.5 [1.79 to 8.99] | 3.55 [2.45 to 11.26]

7. Secondary Outcome: Change in Milk Skin Prick Test Responses
Description: Change in milk skin prick test responses measured as a change in wheal size in millimeters.
Time Frame: Baseline and up to year 2
Population: For change from baseline to year 1, 1 participant dropped out in each group so SPT results only were available for 14 participants in each group. 4 participants dropped out in year 2 so SPT results was available for 12 in each group for change from baseline to year 2.
Measure: Median (95% Confidence Interval); unit: millimeters
Arm/Group | Baked Milk Immunotherapy | Placebo
Number analyzed (Participants) | 14 | 14
millimeters
  Change from baseline to year 1 | -2.5 [-10 to 3] | 3.5 [-2.16 to 14.99]
  Change from baseline to 2 years: number analyzed (Participants) | 12 | 12
  Change from baseline to 2 years | -4 [-7.79 to 1.79] | 1.5 [-6.47 to 10]

8. Secondary Outcome: Change in Quality of Life as Assessed by the Food Allergy Questionnaire
Description: The food allergy questionnaire has an overall score range of 0-6 with 6 indicating the worst quality of life.
Time Frame: Baseline and up to year 2
Population: For change from baseline to year 1, 1 participant dropped out in each group so questionnaire results only were available for 14 participants in each group. 4 participants dropped out in year 2 so questionnaire results was available for 12 in each group for change from baseline to year 2.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baked Milk Immunotherapy | Placebo
Number analyzed (Participants) | 14 | 14
score on a scale
  change from baseline to 1 year | 0.04 (0.79) | 0.37 (1.08)
  change from baseline to 2 years: number analyzed (Participants) | 12 | 12
  change from baseline to 2 years | -0.07 (0.94) | -0.3 (1.16)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse events were recorded by body system affected.
Arm/Group | Baked Milk Immunotherapy | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 3/15
Other Adverse Events (participants affected / at risk) | 15/15 | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baked Milk Immunotherapy (N=15) | Placebo (N=15)
Hospitalization - asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2 (2)
Hospitalization - mental health (Psychiatric disorders) | 0 | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Baked Milk Immunotherapy (N=15) | Placebo (N=15)
Oropharyngeal symptoms (General disorders) | 14 | 8
Cutaneous symptoms (Skin and subcutaneous tissue disorders) | 14 | 12
Gastrointestinal symptoms (Gastrointestinal disorders) | 15 | 14
Lower respiratory tract symptoms (Respiratory, thoracic and mediastinal disorders) | 12 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-09): https://cdn.clinicaltrials.gov/large-docs/30/NCT03462030/Prot_SAP_000.pdf